CLINICAL TRIAL: NCT01298947
Title: Photoablative Atherectomy Followed by a Paclitaxel-Coated Balloon to Inhibit Restenosis in Instent Femoro-popliteal Obstructions
Acronym: PHOTOPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Herz-Zentrums Bad Krozingen (Other)
Responsible Party: Prof. Dr. Thomas Zeller, Herz-Zentrum Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHOTOPAC
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Restenosis
Keywords: Photoablative Atherectomy; Paclitaxel-Coated Balloon; Instent Femoro-popliteal Obstructions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser atherectomy and drug-coated balloon (Active Comparator): Laser atherectomy and Paclitaxel-coated balloon angioplasty in treatment of instent lesions of femoropopliteal arteries
  Interventions: Device: Laser Atherectomy (Spectranetics CE marked peripheral laser atherectomy catheters (including Turbo Elite®), Turbo-Booster® and Turbo Tandem™ Systems
- Drug eluting Ballon PTA (Active Comparator): Paclitaxel-coated balloon angioplasty
  Interventions: Device: Laser Atherectomy (Spectranetics CE marked peripheral laser atherectomy catheters (including Turbo Elite®), Turbo-Booster® and Turbo Tandem™ Systems

INTERVENTIONS:
Device: Laser Atherectomy (Spectranetics CE marked peripheral laser atherectomy catheters (including Turbo Elite®), Turbo-Booster® and Turbo Tandem™ Systems — comparing the use of a Paclitaxel-eluting angioplasty balloon (PTX PTA) with initial photoablation to the use of PTX PTA alone in the treatment of instent lesions in femoropopliteal arteries

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of preparing a vessel with photoablation with Spectranetics CVX-300® Excimer laser and laser catheters prior to local Paclitaxel delivery compared to local Paclitaxel delivery without initial photoablation

DETAILED DESCRIPTION:
This is a prospective, two-arm randomized study. The control cohort (PTX PTA group, Admiral Inpact or Pacific Inpact, Medtronic-Invatec) will be treated with a PTX-coated PTA balloon. The experimental cohort (Laser+PTX PTA group) will be treated with photoablative atherectomy followed by a PTX-coated PTA balloon. Subjects meeting the definitions of Rutherford Clinical Categories 1 to 5 with instent lesions located in superficial femoral artery and the popliteal artery above the knee joint are eligible for enrollment.

The purpose of this feasibility study is to evaluate the safety and effectiveness of preparing an instent lesion with photoablative atherectomy prior to local Paclitaxel delivery compared to local Paclitaxel delivery without initial photoablative atherectomy.

Primary Outcome:

Target Lesion Percent Diameter Stenosis (%DS) at 1 Year defined as the narrowest point of the target lesion divided by the estimated native vessel diameter at that location as determined by the ACL.

Secondary Outcomes:

The following secondary outcomes will be summarized in this study.

1. Procedural Success: Defined as ≤ 30% residual stenosis following the procedure at the target lesion, without periprocedural complications, as determined by the ACL.
2. Major Adverse Event Rate at 30 Days and 1 Year: Defined as major unplanned amputation of the treated limb, all-cause mortality within 1 year of the index procedure or clinically-driven target vessel revascularization within 30 days of the index procedure.
3. Improvement in WIQ Score at 6 Months and 1 Year: Defined as an increase in Walking Impairment Questionnaire (WIQ) score at 6 months and 1 year compared to baseline.
4. Improvement in EQ-5D Score at 6 Months and 1 Year: Defined as an increase in the EQ-5D questionnaire score at 6 months and 1 year compared to baseline.
5. Improvement in Rutherford Clinical Category at 6 Months and 1 Year: Defined as an improvement in clinical status indicated by a decrease of one or more in Rutherford Clinical Category at 6 months and 1 year compared to baseline, that is attributable to the target limb (in cases of bilateral disease).
6. Improvement in Ankle-Brachial Index at 6 Months and 1 Year: Defined as an increase in the ankle-brachial index (ABI) at 6 months and 1 year compared to baseline in subjects with compressible arteries and baseline ABI < 0.9.
7. Clinically-Driven Target Lesion Revascularization (TLR) at 6 Months and 1 Year. Defined as any reintervention or artery bypass graft surgery involving the target lesion in which the subject has ≥ 50% diameter stenosis in the presence of recurrent symptoms (i.e. claudication) or ≥ 70% stenosis without any symptoms (i.e. decreased ABI).
8. Patency Rate (Peak Systolic Velocity ≤ 3.5) at 6 & 12 Months: Defined by duplex ultrasound core lab measurement of peak systolic velocity (PSV) ratio ≤ 3.5 at the target lesion with no clinically-driven reintervention within the target lesion.
9. Alternative Patency Rate (Peak Systolic Velocity ≤ 2.4) at 6 & 12 Months: Defined by duplex ultrasound core lab measurement of peak systolic velocity (PSV) ratio ≤ 2.4 at the target lesion with no clinically-driven reintervention within the target lesion.
10. Minimum Lumen Diameter at 1 Year: Determined by angiographic assessment of the target lesion at 1 year by the ACL.
11. Net Lumen Gain at 1 Year: Defined as the difference between the target lesion MLD at baseline and 1 year following the index procedure per angiographic assessment determined by the ACL.
12. Patency Rate at 1 Year: Defined as ≤ 70% stenosis per angiography as determined by the ACL.
13. Secondary Patency Rate at 1 Year: Defined as ≤ 70% stenosis per angiography as determined by the ACL, maintained by repeat percutaneous intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all of the following general inclusion criteria.

  1. Has a Rutherford Clinical Category Score of 1 - 5.
  2. Is willing and capable of complying with all follow-up evaluations at the specified times.
  3. Is ≥ 18 years old.
  4. Provides written informed consent prior to study specific procedures.

Exclusion Criteria:

* The subject must not meet any of the following general exclusion criteria.

  1. Has contraindications listed in any study device IFUs.
  2. Has a contraindication or known untreated allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs or any other drug anticipated to be used.
  3. Has a hypersensitivity to contrast material that cannot be adequately pretreated.
  4. Has known hypersensitivity to treatment device materials including Paclitaxel. Has known uncontrollable hypercoagulable condition, or refuses blood transfusion.

  6. Has life expectancy of less than 12 months. 7. Is pregnant, of childbearing potential not taking adequate contraceptives, or nursing.

  8. Has surgical or endovascular procedure of the target vessel within 14 days prior to the index procedure.

  9. Has any planned surgical intervention (requiring hospitalization) or endovascular procedure within 30 days after the index procedure.

  10. Is currently participating in an investigational drug or another device study that may clinically interfere with the study outcomes.

  11. Any co-morbid condition that in the judgment of the physician precludes safe percutaneous intervention.

  12. Has had a previous peripheral bypass affecting the target vessel. 13. Has chronic renal insufficiency with creatinine > 2.5 mg/L (except patients under chronic renal replacement therapy).

  14. Is unable or unwilling to receive dual anti-platelet therapy. 15. Equipment is unavailable to fulfill study treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Percent Stenosis | at 1 Year
  Target Lesion Percent Stenosis at 1 Year: Defined as the narrowest point of the target lesion divided by the estimated native vessel diameter at that location as determined by the angiographic core lab.

SECONDARY OUTCOMES:
Procedural Success | at 1 year
  Defined as ≤ 30% residual stenosis following the procedure at the target lesion, without periprocedural complications, as determined by the angiographic core lab.
  Major Adverse Event Rate at 30 Days and 1 Year: Defined as, major unplanned amputation of the treated limb, all-cause mortality within 1 year of the index procedure or clinically-driven target vessel revascularization within 30 days and 1 year of the index procedure.